CLINICAL TRIAL: NCT03257540
Title: Prospective Clinical Evaluation of Early Weight-Bearing After Lapidus Arthrodesis Using the Phantom™ Intramedullary Nail
Brief Title: Early Weight-Bearing After Lapidus Arthrodesis
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: P30-SP-0001
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Arthrodesis; Bunion; Hallux Valgus
Keywords: bunion; early weight-bearing; Lapidus; arthrodesis; intramedullary nail; Hallux Valgus
MeSH Terms: conditions — Ankylosis; Bunion; Hallux Valgus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Small Bone Intramedullary Nail: All study participants
  Interventions: Device: Small Bone Intramedullary Nail

INTERVENTIONS:
Device: Small Bone Intramedullary Nail — Patients undergoing a Lapidus Arthrodesis procedure for hallux valgus correction who are receiving a Phantom Small Bone Intramedullary nail will begin weight-bearing at 2 weeks and follow a pre-determined post-operative protocol.
  Other Names: Phantom Small Bone Intramedullary Nail - Lapidus

SUMMARY:
The goal of this research study is to determine if union rates are affected by early weight-bearing after Lapidus Arthrodesis using the Phantom™ Intramedullary Nail.

The study hypothesis is that the union rate for those who undergo a Lapidus Arthrodesis procedure with the Phantom™ Intramedullary Nail and participate in an early weight-bearing protocol will be non-inferior to union rates previously published for this procedure.

DETAILED DESCRIPTION:
Each subject will undergo a Lapidus Arthrodesis which entails cartilage removal from the 1st TMT joint, subchondral bone preparation, deformity correction, temporary fixation and permanent fixation with the Phantom™ Intramedullary Nail. The Phantom™ Intramedullary Nail is inserted by drilling a hole for the nail at a specified location using instrumentation and a targeting guide. The nail is inserted into the drill hole and is fixated to the medial cuneiform and 1st metatarsal using three threaded pegs and a locking screw.

A subchondral drill and chisel are provided in the system with the Lapidus Nail. Subchondral drilling and feathering of the subchondral bone with a chisel are standard ways to prepare the subchondral bone and elicit bleeding bone prior to arthrodesis. Use of this instrumentation is encouraged for this study to ensure that proper bone preparation is performed for arthrodesis. A torque indicating driver is also encouraged to be used for this procedure to help guide the surgeon to appropriate compression to apply across the joint. Alternatively, a standard driver and handle can be used with two-finger tightness when compressing the joint to achieve a similar effect.

Traditionally, it is common for people who undergo a Lapidus Arthrodesis to be non-weight-bearing for 6-8 Weeks following the surgical procedure. This time allows the bones to properly fuse together. During this 6-8 week period, people can be limited in the typical day-to-day activities they participate in, such as walking, shopping and working.

The Phantom™ Intramedullary Nail may allow subjects to bear weight earlier than traditional procedures without negatively effecting fusion. By allowing people to bear weight earlier than traditional methods, it is possible that people will have the opportunity to resume typical day-to-day activities faster than usual.

The study in question will investigate the Phantom™ Intramedullary Nail with the following early weight-bearing protocol (see "Post-Operative Protocol for Study Participant" below).

The study preference is that subjects are placed in a splint from 0-2 Weeks. However, a cast may be substituted according to surgeon preference. No casts are permitted beyond 2 Weeks, unless deemed as a medical necessity in which case the subject would no longer follow the early weight-bearing protocol.

The study preference is that subject will be placed in a walking boot at 2 Weeks. However, an immobilizing shoe may be substituted according to surgeon preference.

Post-Operative Protocol for Study Participant

Activity Level Definitions:

Sedentary: Most activities are done seated or lying down. Surgically repaired foot should be raised when in seated or reclined position. Standing limited to less than 15 minutes per hour. Moving is limited to necessary activities such as going to the bathroom or food preparation.

Light Activity: Standing limited to less than 30 minutes per hour. Movement is mostly limited to in-home movement such as folding laundry or wiping counters. Short time periods of movement to leave the house can be performed for necessary activities (such as the grocery store), but should be limited to less than 30 minutes of standing time.

Moderate Activity: No limits on standing. Walking limited to 45 minute time periods no more than 3 times per day. No running, jumping or heavy lifting (more than 25 pounds).

Heavy Activity: No limits on walking, running and jumping. No lifting limits.

0-2 Weeks After Surgery:

* Footwear: You will have a splint (or cast) on your surgically repaired foot/leg. The splint (or cast) should not be removed. You will wear a comfortable shoe on the other foot.
* Weight-Bearing: Do not put any weight on your surgically repaired foot.
* Mobility Aid: You will use a walking aid such as crutches, rolling knee scooter or wheelchair to keep all weight off of your surgically repaired foot.
* Range of Motion Exercises: None.
* Activity level: Sedentary after surgery working up to light activity over two Weeks (restarting activities of daily living without putting weight on your foot).

2-6 Weeks After Surgery:

* Footwear: A restrictive boot (or shoe) will be given to you by your doctor. This should not be removed other than for range of motion exercises and bathing (seated). Wear a comfortable shoe on the other foot.
* Weight-Bearing: Put weight on your foot as you can tolerate in the restrictive boot (or shoe). Do not walk without the restrictive boot (or shoe).
* Mobility Aid: If possible, no walking aid should be used. If needed for pain, use a walking aid as necessary.
* Range of Motion Exercises: You will do range of motion exercises without the restrictive boot (or shoe) with no weight on your foot, as instructed by your doctor.
* Activity level: Light activity with restrictive boot (or shoe). 6 Weeks-3 Months After Surgery:
* Footwear: You will wear a restrictive boot (or shoe) working up to supportive shoe (preferably a lace-up or Velcro shoe including sneakers, running shoes, work boots or soft leather shoes without a heel) by 8 Weeks after your surgery.
* Weight-Bearing: Put weight on your foot as you can tolerate. Barefoot walking is not encouraged.
* Mobility Aid: No help from crutches, scooter, or wheelchair.
* Range of Motion Exercises: You will do range of motion exercises as instructed by your doctor.
* Activity level: Light activity working up to moderate activity (low impact) as you can tolerate.

3-6 Months After Surgery:

* Footwear: At Month 3-4, move from a supportive shoe to footwear of your choice, as you can tolerate.
* Weight-Bearing: Put weight on your foot as you can tolerate.
* Mobility Aid: No help from crutches, scooter, or wheelchair.
* Activity level: Moderate activity for 3-4 Months post-operative, slowly moving into heavy activity as you can tolerate after Month 4.

  6 Months - 2 Years After Surgery:
* Footwear: You have no restrictions on footwear.
* Weight-Bearing: Put weight on your foot as you can tolerate.
* Mobility Aid: No help from crutches, scooter, or wheelchair.
* Activity Level: No activity limits.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age with closed physeal plates at the time of screening.
* The intermetatarsal angle is greater than or equal to 10 degrees.
* The hallux valgus angle is greater than or equal to 25 degrees.
* The subject has foot pain/discomfort on the foot in question.
* The subject has activity limitations due to the foot in question.
* The subject agrees to comply with the requirements of the study and complete the study measures.
* The subject is willing and able to provide written informed consent.

Exclusion Criteria:

* The subject is pregnant.
* The subject is a current smoker.
* The subject has been clinically diagnosed with diabetes.
* The subject has been clinically diagnosed with peripheral neuropathy.
* The subject had been previously sensitized to titanium.
* The subject currently takes oral steroids or rheumatoid biologics.
* The subject has had previous surgery for hallux valgus on operative side.
* The subject has insufficient quantity or quality of bone to permit stabilization, conditions that retard healing (not including pathological fractures) and conditions causing poor blood supply such as peripheral vascular disease.
* The subject has a history of delayed or non-union for fracture or joint.
* The subject has an active, suspected or latent infection in the affected area.
* The subject will require a structural graft in the 1st TMT joint.
* The subject is scheduled to undergo a concomitant 2nd tarsometatarsal joint arthrodesis procedure.
* The subject is scheduled to undergo a same-day bilateral procedure.
* The subject cannot be scheduled for surgery within 3 months of the pre-operative exam.
* The subject has previously been enrolled into this study for a contralateral procedure.
* The subject is actively involved with a Workman's Compensation case.
* The subject is not expected to complete the study according to the investigation plan.
* The subject has been deemed physiologically or psychologically inadequate by the enrolling physician.
* The subject is: a prisoner, unable to understand what participation in the study entails, mentally incompetent, a known abuser of alcohol and/or drugs or anticipated to be non-compliant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults age 18 and older with a painful bunion deformity. The most common age demographic to have surgery for hallux valgus correction is age 50-59. Additionally, the prevalence of hallux valgus in females is greater than males, so a higher percentage of female subjects seeking treatment is likely to be expected.
  This population is suitable for the purpose of the investigation, as groups most likely to seek treatment (surgical) for hallux valgus correction will be represented in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical/radiographic healing | 6 months
  Evaluate clinical/radiographic healing (union vs. non-union) after a Lapidus arthrodesis procedure at 6 months following a surgery using the Phantom Intramedullary nail with early weightbearing at 2 weeks.

SECONDARY OUTCOMES:
Clinical complications | 24 Months
  Complications due to the procedure or post-operative protocol or health conditions that could affect other outcome measures
Time to full weight-bearing | 0 to 12 months
  The amount of time needed for a participant to become fully weight-bearing after the Lapidus surgery.
Change in radiographic angular/positional alignment before and after the Lapidus procedure | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  Hallux Abductus Angle Intermetatarsal Angle First Metatarsal Declination Angle Distal Metatarsal Articular Angle Sesamoid Position
Change in VAS Pain Score across multiple time points | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  Patient reported pain
Change in AOFAS Forefoot/Hallux Valgus Score across multiple time points | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  Clinical score
Change in PROMIS Mobility Score across multiple time points | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  Patient reported mobility assessment, Item Bank v2.0
Change in PROMIS Pain Interference Score across multiple time points | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  Patient reported pain interference assessment, Item Bank v1.0, SF 6a
Change in PROMIS Pain Intensity Score across multiple time points | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  Patient reported pain intensity assessment, Item Bank v1.0, SF 3a
Evaluate time to return to work post-operatively while noting labor classification | 0 to 24 months
  sedentary, light labor, medium labor, heavy labor, very heavy labor
Evaluate time to return to full duty work post-operatively while noting labor classification | 0 to 24 months
  sedentary, light labor, medium labor, heavy labor, very heavy labor
Change in Range of Motion across multiple time points | Pre-operatively, 2 Weeks, 6 Weeks, 12 Weeks, 6 Months, 12 Months, 24 Months
  1st MTP Dorsiflexion
  1st MTP Plantarflexion Ankle Dorsiflexion Ankle Plantarflexion

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Redwood Orthopaedic Surgery Associates, Santa Rosa, California
  - Orthopaedic & Spine Center of the Rockies, Fort Collins, Colorado
  - Orthopedic Center of Palm Beach County, Atlantis, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casaburi R, Porszasz J, Hecht A, Tiep B, Albert RK, Anthonisen NR, Bailey WC, Connett JE, Cooper JA Jr, Criner GJ, Curtis J, Dransfield M, Lazarus SC, Make B, Martinez FJ, McEvoy C, Niewoehner DE, Reilly JJ, Scanlon P, Scharf SM, Sciurba FC, Woodruff P; COPD Clinical Research Network. Influence of lightweight ambulatory oxygen on oxygen use and activity patterns of COPD patients receiving long-term oxygen therapy. COPD. 2012 Feb;9(1):3-11. doi: 10.3109/15412555.2011.630048. PMID 22292592